CLINICAL TRIAL: NCT06446648
Title: Impact of Intraoperative ICG Use During Robotic-Assisted Radical Prostatectomy on Functional Outcomes
Brief Title: Impact of Intraoperative ICG on Functional Outc in RARP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, David Inkoo Lee, Professor of Clinical Urology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4845; UCI 23-137 (Other: UCI CFCCC)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOC group (No Intervention): Robot-Assisted Radical Prostatectomy will be performed as a standard procedure.
- ICG group (Experimental): Robot-Assisted Radical Prostatectomy using ICG
  Interventions: Drug: ICG

INTERVENTIONS:
Drug: ICG — Administer an IV ICG injection intraoperatively, using the optimal dosage and timing defined in the second phase of the study. Utilize the newly developed 3D vascular map for visualization of the arteries before and after prostate resection.
  Other Names: Indocyanine Green
  Arms: ICG group

SUMMARY:
This is a pilot, 3 phases open-label feasibility study with the 3rd phase consisting of randomized 2-arm intervention trial, to assess the systematic use of indocyanine green (ICG) in subjects with prostate adenocarcinoma during robot-assisted radical prostatectomy and its impact on sexual function outcomes at 12 months postoperatively.

DETAILED DESCRIPTION:
The first phase of this study will involve performing 50 cases of nerve-sparing RARP on patients who are good candidates for nerve sparing. During these procedures, we will record the location and size of arteries encountered to create a detailed 3D map of the surgical arterial vasculature.

In the second phase, we will recruit another 50 patients. These patients will receive an IV injection of ICG before encountering the arteries to visualize them prior to resection. This phase will determine the optimal dosage and timing for the IV ICG injection.

The third phase will utilize the dosage and timing defined in the second phase. This phase will be a randomized trial involving 300 patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must be ≥18 years old, male, and sexually active.
* 2. Histologically/pathologically confirmed localized prostate adenocarcinoma.
* 3. Most recent preoperative Sexual Health Inventory for Men (SHIM) score ≥16.
* 4. Subjects who are candidates for good nerve sparing preoperatively determined by the investigator by assessing imaging findings.
* 5. Ability to read, write and understand and willingness to sign a written informed consent.
* 6. Subjects must pass medical clearance from primary care provider and cardiologist, if applicable.
* 7. Subject must be determined to be medical fit for RARP by the investigator.

Exclusion Criteria:

* 1. No locally advanced or metastatic prostate adenocarcinoma.
* 2. Preoperative diagnosis of erectile dysfunction with any use of invasive interventions such as intrapenile injections and intrapenile prosthesis implants. Oral interventions are acceptable and are not exclusionary.
* 3. Received neoadjuvant treatment for high-risk prostate cancer or received prior focal treatment of the prostate or prior definitive radiotherapy.
* 4. History of allergic reactions attributed to ICG.
* 5. Subjects who are preoperatively not foreseen as ideal candidates for nerve sparing interventions by the investigator.
* 6. Subjects who are unable to comply with study and follow-up procedures as judged by the investigator.
* 7. Subjects who are illiterate.
* 8. Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interpretation of outcomes, including active opportunistic infections or advanced (severe) infections, or uncontrolled diabetes.
* 9. Any other disease, metabolic disorder, or abnormal finding upon physical examination or laboratory examination that makes the subject unsuitable for receiving the intervention, affects the interpretation of study outcomes, or poses risks to subject safety, as determined by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Continence Rate at 3 month Post-surgery | 3 months
  Number of patients who report using no pads or only 1 security pad per day at 3-month post-surgery.

SECONDARY OUTCOMES:
Patient Reported Continence and Sexual Functions | 12 months
  Subjects will complete the investigator-developed, "Follow Up Continence And Sexual Function" questionnaires. This questionnaire includes questions typically asked in Sexual Health Inventory for Men (SHIM) and International Prostate Symptom Score (IPSS) surveys and assesses postoperative functional outcomes such as urinary continence/leakage, daily pad usage, sexual function such as percentage fullness of erection and postoperative.
  The scales used are the:
  * Sexual Health Inventory for Men (SHIM), with a minimum value of 1 and a maximum value of 25. A higher score indicates a better outcome, and
  * the Internatioanl Prostate Symptom Score (IPSS), with a minimum value of 0 and a maximum of 35. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No